CLINICAL TRIAL: NCT00807742
Title: Contingent Vouchers for Smoking in Substance Abusers as Adjunct to Nicotine Patch
Brief Title: Contingency Management for Smoking in Substance Abusers
Acronym: SCMSUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Damaris J. Rohsenow, Ph.D., Professor (Research): Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA023995-01 (NIH); R01DA023995 (NIH)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Substance Abuse
Keywords: Contingency management for smoking for substance abusers; Contingency reinforcement for smoking abstinence; Contingency Management; Noncontingent Reinforcement
MeSH Terms: conditions — Substance-Related Disorders | interventions — Nicotine Replacement Therapy; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (CM) (Experimental): Condition provides contingent monetary reinforcement for smoking reductions (first 5 days) then for smoking abstinence (subsequent 14 days). Expired carbon monoxide (CO) levels will be the basis for determining reductions and abstinence.
  Interventions: Drug: Nicotine Replacement Treatment (NRT); Behavioral: Brief Advice; Behavioral: Contingency Management
- Noncontingent Reinforcement (NR) (Active Comparator): Controls for effects of receiving payments, providing daily breath samples for CO level, and degree of interaction between patient and research staff. NR will allow them to earn an amount which is matched in amount to the expected average earned in CM contingent only on providing breath samples independent of the CO level attained.
  Interventions: Drug: Nicotine Replacement Treatment (NRT); Behavioral: Brief Advice; Behavioral: Non-Contingent Reinforcement

INTERVENTIONS:
Drug: Nicotine Replacement Treatment (NRT) — Nicoderm CQ nicotine skin patch: 21mg patch for 4 weeks, 14mg patch for 2 weeks, 7mg patch for 2 weeks. This is supplemental intervention provided to all.
  Other Names: Nicoderm CQ skin patch; Nicotine replacement therapy
Behavioral: Brief Advice — Brief Advice (BA): Patients will receive four sessions of a manualized brief intervention based on NCI guidelines (Manley et al., 1991; Hollis et al., 1993) as modified for sobriety settings. This simple counseling has five components: (1) Assess smoking and initial interest in cessation; (2) Advise the patient to quit smoking; (3) Assist the patient in quitting; (4) Assess interest in quitting; and (5) Arrange booster sessions. This supplemental information is provided to all.
  Other Names: Smoking counseling
Behavioral: Contingency Management — Condition provides contingent monetary reinforcement for smoking reductions (first 5 days) then for smoking abstinence (subsequent 14 days). Expired carbon monoxide (CO) levels will be the basis for determining reductions and abstinence.
  Arms: Contingency Management (CM)
Behavioral: Non-Contingent Reinforcement — Controls for effects of receiving payments, providing daily breath samples for CO level, and degree of interaction between patient and research staff. NR will allow them to earn an amount which is matched in amount to the expected average earned in CM contingent only on providing breath samples independent of the CO level attained.
  Arms: Noncontingent Reinforcement (NR)

SUMMARY:
The aim of this study is to determine whether contingent reinforcement for smoking abstinence, compared to noncontingent reinforcement, increases the effectiveness of brief counseling and nicotine replacement on smoking abstinence of substance abusers in residential treatment.

DETAILED DESCRIPTION:
Substance abusers have a high prevalence and rate of smoking with little success in quitting, so stronger approaches are needed to encourage attempts to quit smoking.

The aim of this study is to determine whether contingent reinforcement for smoking abstinence (CM), compared to noncontingent reinforcement (NR), increases the effectiveness of brief counseling and nicotine replacement on smoking abstinence of substance abusers in residential treatment. The proposed study will be a 2-group design in which up to 274 substance abusers who smoke 10 or more cigarettes per day receive brief advice (4 sessions) and nicotine replacement (NRT) (8 weeks), and are randomized to 19 days of CM for smoking vs. a matched NR condition. The brief advice is adapted slightly for sobriety settings. Point-prevalence abstinence will be assessed at 1, 3, 6 and 12 months after starting treatment. Secondary aims evaluate effects of CM on substance use outcomes and potential mediators of effects on outcome, including within-treatment abstinence, motivation level and tolerance for smoking discomfort.

The significance is to add knowledge about the most effective ways to maximize smoking cessation among substance abusers, important given that no methods are known to work with this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of substance abuse or dependence by DSM-IV criteria
* in residential treatment at one particular agency
* currently smoking at least 10 cigarettes per day for the past 6 months

Exclusion Criteria:

* hallucinating or delusional or marked organic impairment (to the point of impairing ability to understand informed consent) according to medical records
* current use of nicotine replacement therapy, Zyban, or any other smoking cessation treatment
* medical exclusions for NRT: pregnant or nursing; treatment in the last 3 months for unstable angina, severe congestive heart failure, uncontrolled hypertension; lung cancer; supplemental oxygen; history of adverse reactions to NRT; allergies to adhesive; or any severe skin disease that requires treatment (e.g., psoriasis or eczema).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2008-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damaris Rohsenow, Ph.D., Principal Investigator — Brown University; Rosemarie Martin, Ph.D., Study Director — Brown University
Locations (1):
- Brown University, Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Rohsenow DJ, Monti PM, Colby SM, Martin RA. Brief interventions for smoking cessation in alcoholic smokers. Alcohol Clin Exp Res. 2002 Dec;26(12):1950-1. doi: 10.1097/01.ALC.0000041006.59547.9A. No abstract available. PMID 12500132
- [Background] Rohsenow DJ, Martin RA, Tidey JW, Colby SM, Monti PM. Treating Smokers in Substance Treatment With Contingent Vouchers, Nicotine Replacement and Brief Advice Adapted for Sobriety Settings. J Subst Abuse Treat. 2017 Jan;72:72-79. doi: 10.1016/j.jsat.2016.08.012. Epub 2016 Aug 18. PMID 27658756
- [Result] Mackillop J, Murphy CM, Martin RA, Stojek M, Tidey JW, Colby SM, Rohsenow DJ. Predictive Validity of a Cigarette Purchase Task in a Randomized Controlled Trial of Contingent Vouchers for Smoking in Individuals With Substance Use Disorders. Nicotine Tob Res. 2016 May;18(5):531-7. doi: 10.1093/ntr/ntv233. Epub 2015 Oct 24. PMID 26498173

RESULTS

PARTICIPANT FLOW:
Groups:
- Contingency Management (CM): Condition provides contingent monetary reinforcement for smoking reductions (first 5 days) then for smoking abstinence (subsequent 14 days). Expired carbon monoxide (CO) levels will be the basis for determining reductions and abstinence.
  Nicotine Replacement Treatment (NRT): Nicoderm CQ nicotine skin patch: 21mg patch for 4 weeks, then 14mg patch for 2 weeks and 7mg patch for 2 weeks. This is supplemental intervention provided to all.
  Brief Advice: Brief Advice (BA): Patients receive four sessions of a manualized brief intervention based on NCI guidelines (Manley et al., 1991; Hollis et al., 1993) as modified for sobriety settings. This simple counseling has five components: (1) Assess smoking and initial interest in cessation; (2) Advise the patient to quit smoking; (3) Assist the patient in quitting; (4) Assess interest in quitting; and (5) Arrange booster sessions. This supplemental information is provided to all.
- Noncontingent Reinforcement (NR): Controls for receiving payments, providing daily breath samples for CO level, and interaction between patient and research staff. NR allows them to earn an amount which is matched in amount to the expected average earned in CM contingent only on providing breath samples independent of the CO level.
  Nicotine Replacement Treatment (NRT): Nicoderm CQ nicotine skin patch: 21mg patch for 4 weeks, 14mg patch for 2 weeks, 7mg patch for 2 weeks. This is supplemental intervention provided to all.
  Brief Advice: Brief Advice (BA): Patients receive four sessions of a manualized brief intervention based on NCI guidelines (Manley et al., 1991; Hollis et al., 1993) as modified for sobriety settings. This simple counseling has five components: (1) Assess smoking and initial interest in cessation; (2) Advise the patient to quit smoking; (3) Assist the patient in quitting; (4) Assess interest in quitting; and (5) Arrange booster sessions. This supplemental information is provided to all.
Period: Overall Study
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Started | 172 | 168
Completed | 126 | 114
Not Completed | 46 | 54
Not completed — Death | 9 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 35 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR) | Total
Number analyzed (Participants) | 172 | 168 | 340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 172 | 168 | 340
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.87 (10.14) | 37.28 (9.95) | 37.58 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 52 | 111
  Male | 113 | 116 | 229
Region of Enrollment [Number; unit: participants]
  United States | 172 | 168 | 340

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Smoking Abstinent in Past 7 Days
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 1-month follow-up
Population: "Intent to Treat" Note: People who were lost were counted as smoked.
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 172 | 168
participants | 16 | 13
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .606, Chi-squared; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.57 to 2.63]

2. Primary Outcome: Number of Participants Smoking Abstinent in Past 7 Days
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 3-month follow up
Population: "Intent to Treat" Note: People who were lost were counted as smoked. 3 participants died before 3 month follow up were coded as missing.
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 170 | 167
participants | 9 | 5
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .290, Chi-squared; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.57 to 2.63]

3. Primary Outcome: Number of Participants Smoking Abstinent in Past 7 Days
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 6-month follow up
Population: "Intent to Treat" Note: People who were lost were counted as smoked. 5 participants died before 6 month follow up were coded as missing.
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 168 | 167
participants | 6 | 3
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .32, Chi-squared; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.49 to 8.23]

4. Primary Outcome: Number of Participants Smoking Abstinent in Past 7 Days
Description: 7 -day smoking cessation confirmed by expired alveolar CO levels of < 10 ppm or salivary cotinine < 16 ng/ml.
Time Frame: 12-month follow up
Population: "Intent to Treat" Note: People who were lost were counted as smoked. 11 participants died before 12 month follow up were coded as missing.
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 163 | 166
participants | 6 | 3
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .298, Chi-squared; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.51 to 8.45]

5. Primary Outcome: Average Number of Cigarettes Per Day
Time Frame: 1-month follow up
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 172 | 168
cigarettes | 5.28 (5.49) | 7.98 (5.49)
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p < .001, t-test, 2 sided; Effect Size d = -0.49, 95% CI 2-sided [-0.71 to -0.27]

6. Primary Outcome: Average Number of Cigarettes Per Day
Time Frame: 3-month follow up
Population: Outcome data available for 291 participants who completed 3 month follow up. 3 participants died and 46 were lost to follow up before 3 month follow up.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 148 | 143
cigarettes | 8.84 (7.57) | 9.89 (6.19)
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .199, t-test, 2 sided; Effect Size d = -0.15, 95% CI 2-sided [-0.38 to 0.08]

7. Primary Outcome: Average Number of Cigarettes Per Day
Description: Timeline Followback interview assessing number of cigarettes on each day of each 3-month reporting period
Time Frame: 6-month follow up
Population: Outcome data available for 268 participants who completed 6 month follow up. 5 participants died and 67 were lost to follow up before 6 month follow up.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 138 | 130
cigarettes | 10.87 (8.05) | 12.18 (6.59)
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .148, t-test, 2 sided; Effect Size d = -0.12, 95% CI 2-sided [-.57 to 0.33]

8. Primary Outcome: Average Number of Cigarettes Per Day
Time Frame: 12-month follow up
Population: Outcome data available for 240 participants who completed 12 month follow up. 11 participants died and 89 were lost to follow up before 12 month follow up.
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 126 | 114
cigarettes | 11.67 (7.70) | 12.78 (7.23)
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .249, t-test, 2 sided; Effect Size d = -0.15, 95% CI 2-sided [-0.40 to 0.11]

9. Primary Outcome: Number of Participants With Relapse to Any Heavy Drinking
Description: Heavy drinking = 6 or more drinks for men; 5 or more drinks for women
Time Frame: 1-month follow up
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 172 | 168
participants | 12 | 8
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = 0.402, Chi-squared; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.59 to 3.72]

10. Primary Outcome: Number of Participants With Relapse to Any Heavy Drinking
Description: Heavy drinking = 6 or more drinks for men; 5 or more drinks for women
Time Frame: 3-month follow up
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 148 | 143
participants | 23 | 24
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .772, Chi-squared; Odds Ratio (OR) = .91, 95% CI 2-sided [0.49 to 1.70]

11. Primary Outcome: Number of Participants With Relapse to Any Heavy Drinking
Description: Heavy drinking = 6 or more drinks for men; 5 or more drinks for women
Time Frame: 6-month follow up
Population: Outcome data available for 268 participants who completed 3 month follow up. 5 participants died and 67 were lost to follow up before 3 month follow up.
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 138 | 130
participants | 38 | 35
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .910, Chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.60 to 1.77]

12. Primary Outcome: Number of Participants With Relapse to Any Heavy Drinking
Description: Heavy drinking = 6 or more drinks for men; 5 or more drinks for women
Time Frame: 12-month follow up
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 126 | 114
participants | 38 | 36
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .812, Chi-squared; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.54 to 1.62]

13. Primary Outcome: Number of Participants With Relapse to Any Drug Use
Time Frame: 1-month follow up
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 172 | 168
participants | 13 | 16
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .490, Chi-squared; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.36 to 1.65]

14. Primary Outcome: Number of Participants With Relapse to Any Drug Use
Time Frame: 3-month follow up
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 148 | 143
participants | 38 | 32
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .511, Chi-squared; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.67 to 2.06]

15. Primary Outcome: Number of Participants With Relapse to Any Drug Use
Time Frame: 6-month follow up
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 138 | 130
participants | 50 | 42
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .499, Chi-squared; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.72 to 1.97]

16. Primary Outcome: Number of Participants With Relapse to Any Drug Use
Time Frame: 12-month follow up
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 126 | 114
participants | 54 | 50
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority; p = .876, Chi-squared; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.58 to 1.60]

17. Primary Outcome: Percent Smoking Days
Time Frame: 1-month follow up
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 172 | 168
percentage of days | 77.51 (33.02) | 88.33 (25.48)
Statistical Analysis 1: Comparison: Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .001, t-test, 2 sided; Effect Size d = -0.37, 95% CI 2-sided [-0.59 to -0.15]

18. Primary Outcome: Percent Smoking Days
Time Frame: 3-month follow up
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 148 | 143
percentage of days | 82.39 (30.63) | 88.40 (25.48)
Statistical Analysis 1: Comparison: Contingency Management (CM) vs Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .069, t-test, 2 sided; Effect Size d = -0.25, 95% CI 2-sided [-0.46 to 0.02]

19. Primary Outcome: Percent Smoking Days
Time Frame: 6-month follow up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 138 | 130
percentage of days | 88.49 (26.45) | 92.30 (21.91)
Statistical Analysis 1: Comparison: Contingency Management (CM) vs Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .202, t-test, 2 sided; Effect Size d = -0.16, 95% CI 2-sided [-0.40 to 0.08]

20. Primary Outcome: Percent Smoking Days
Time Frame: 12-month follow up
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
Number analyzed (Participants) | 126 | 114
percentage of days | 87.38 (26.62) | 91.53 (22.86)
Statistical Analysis 1: Comparison: Contingency Management (CM) vs Noncontingent Reinforcement (NR); Test type: Superiority or Other; p = .199, t-test, 2 sided; Effect Size d = -0.17, 95% CI 2-sided [-0.42 to 0.09]

ADVERSE EVENTS:
Arm/Group | Contingency Management (CM) | Noncontingent Reinforcement (NR)
All-Cause Mortality (participants affected / at risk) | 9/172 | 2/168
Serious Adverse Events (participants affected / at risk) | 42/172 | 34/168
Other Adverse Events (participants affected / at risk) | 142/172 | 143/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency Management (CM) (N=172) | Noncontingent Reinforcement (NR) (N=168)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Infection (Infections and infestations) | 6 (7) | 4 (4)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Psychiatric (Psychiatric disorders) | 23 (37) | 17 (29)
Medical/Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Nervous System (Nervous system disorders) | 2 (2) | 1 (1)
Renal (Renal and urinary disorders) | 1 (1) | 0 (0)
Social Circumstance (Social circumstances) | 3 (3) | 0 (0)
Vascular (Vascular disorders) | 1 (1) | 1 (1)
Cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Multiple (General disorders) | 0 (0) | 1 (1)
GI (Gastrointestinal disorders) | 0 (0) | 3 (3)
Immune (Immune system disorders) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Contingency Management (CM) (N=172) | Noncontingent Reinforcement (NR) (N=168)
Vivid Dreams/Nightmares (Psychiatric disorders) | 91 | 85
Trouble Sleeping (Psychiatric disorders) | 53 | 58
Skin Irritation (Skin and subcutaneous tissue disorders) | 88 | 86
Tense, Nervous, Anxious (Psychiatric disorders) | 67 | 68
Nausea (Gastrointestinal disorders) | 54 | 59
Headache (Nervous system disorders) | 11 | 18
Dizziness (Ear and labyrinth disorders) | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No